CLINICAL TRIAL: NCT02367664
Title: A Single-centre Phase III Clinical Trial for Vero Cell-derived Inactivated Japanese Encephalitis Vaccine Produced by Shandong Hengye Biotech Co., Ltd. in Healthy Chinese Infants Aged 6-11 Months, Aimed to Evaluate Immunogenicity and Safety
Brief Title: A Clinical Trial for Inactivated Japanese Encephalitis Vaccine in Healthy Chinese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Shandong Hengye Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JSVCT015
Record Dates: First submitted 2015-02-02; First posted 2015-02-20 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Encephalitis
Keywords: Japanese encephalitis; immunogenicity; safety; vaccine
MeSH Terms: conditions — Encephalitis; Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.5ml experimental vaccine on day 0,7 (Experimental): 0.5ml experimental vaccine on day 0,7 and a booster dose 12 months later
  Interventions: Biological: 0.5ml experimental vaccine on day 0,7 Vero cell-derived inactivated Japanese Encephalitis vaccine
- 0.5ml experimental vaccine on day 0,28 (Experimental): 0.5ml experimental vaccine on day 0,28 and a booster dose 12 months later
  Interventions: Biological: 0.5ml experimental vaccine on day 0,28 Vero cell-derived inactivated Japanese Encephalitis vaccine
- 0.5ml active comparator vaccine on day 0,7 (Active Comparator): 0.5ml active comparator vaccine on day 0,7 and a booster dose 12 months later
  Interventions: Biological: 0.5ml active comparator vaccine on day 0,7 inactivated freeze-dried Japanese Encephalitis vaccine(Vero cell)

INTERVENTIONS:
Biological: 0.5ml experimental vaccine on day 0,7 Vero cell-derived inactivated Japanese Encephalitis vaccine — Vero cell-derived inactivated Japanese Encephalitis vaccine produced by Shandong Hengye Biotech Co., Ltd./0.5ml, two doses with 7 days interval, a booster dose 12 months after the first dose
  Arms: 0.5ml experimental vaccine on day 0,7
Biological: 0.5ml experimental vaccine on day 0,28 Vero cell-derived inactivated Japanese Encephalitis vaccine — Vero cell-derived inactivated Japanese Encephalitis vaccine produced by Shandong Hengye Biotech Co., Ltd./0.5ml, two doses with 28 days interval, a booster dose 12 months after the first dose
  Arms: 0.5ml experimental vaccine on day 0,28
Biological: 0.5ml active comparator vaccine on day 0,7 inactivated freeze-dried Japanese Encephalitis vaccine(Vero cell) — inactivated freeze-dried Japanese Encephalitis vaccine(Vero cell) produced by Beijing Tiantan Biological Products Co., Ltd. /0.5ml, two doses with 7 days interval, a booster dose 12 months after the first dose
  Arms: 0.5ml active comparator vaccine on day 0,7

SUMMARY:
Japanese encephalitis (JE) is an acute viral zoonotic disease. Neurologic manifestations of the disease range from subtle changes in behavior to serious problems, including blindness, ataxia, weakness, and movement disorders. The Japanese encephalitis virus (JEV) occurs primarily in Southeast Asian. It is spread by culicine mosquitoes, most often Culex tritaeniorhynchus. Its incubation period is 5 to 15 days.In China, JE epidemic peak season is from June to August and it mainly occurred in children. JE has ranked in top ten infectious diseases according to either incidence or mortality. JE vaccines are used to protect the population especially young children and infants from encephalitis diseases. Live attenuated JE vaccines are now widely used. They are directly produced from attenuated virus which may increase the possibility of virulence reversion. Many developed countries are using purified model inactivated JE vaccine. Therefore, it is an inevitable trend in China to develop a new generation of safer and more effective inactivated vaccine to prevent and control epidemic encephalitis.

DETAILED DESCRIPTION:
Japanese encephalitis (JE) is an acute viral zoonotic disease. Neurologic manifestations of the disease range from subtle changes in behavior to serious problems, including blindness, ataxia, weakness, and movement disorders. The Japanese encephalitis virus (JEV) occurs primarily in Southeast Asian. It is spread by culicine mosquitoes, most often Culex tritaeniorhynchus. Its incubation period is 5 to 15 days. In China, JE epidemic peak season is from June to August and it mainly occurred in children. JE has ranked in top ten infectious diseases according to either incidence or mortality. JE vaccines are used to protect the population especially young children and infants from encephalitis diseases. Live attenuated JE vaccines are now widely used. They are directly produced from attenuated virus which may increase the possibility of virulence reversion. Many developed countries are using purified model inactivated JE vaccine. Therefore, it is an inevitable trend in China to develop a new generation of safer and more effective inactivated vaccine to prevent and control epidemic encephalitis.

In order to evaluate immunogenicity and safety of Vero cell-derived inactivated Japanese Encephalitis vaccine produced by Shandong Hengye Biotech Co., Ltd. a single-centre phase III clinical trial is planned to conduct in healthy infants aged 6-11 months in China.

There will be two immunization programs. 600 healthy infants aged 6-11 months will be randomly assigned (1:1) to receive an experimental vaccine or a positive control vaccine at day 0,7. Another 300 healthy infants aged 6-11 months will be recruited to receive an experimental vaccine at day 0,28. All of them will be received a third dose as booster vaccination 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 6 to 11 months old on the day of inclusion
* Had never received any Japanese Encephalitis vaccine
* Subjects' legal guardians are able to understand and sign the informed consent
* In good general health judged from medical history and clinical examination at the time of inclusion
* Subjects and legal guardians can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Subject who has a medical or family history of any of the following: allergic history, seizure, epilepsy, brain or mental disease
* Subject who is allergic to any ingredient of the vaccine
* Family history of congenital or hereditary immunodeficiency
* Subject with damaged or low immune function which has already been known
* Subject who had a Japanese Encephalitis medical history
* Subject with acute febrile illness or infectious disease
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Thrombocytopenia, blood coagulation disorder or bleeding difficulties with intramuscular injection
* Subject who has serious allergic history
* Subject with other medical history not suitable for vaccination such as fainting during injection or acupuncture treatment
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of any attenuated live vaccine in last 30 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Any acute infection or serious infection needing systemic antibiotics or antiviral treatment in last 7 days
* Any fever with temperature >=38.0°C on axillary setting in last 3 days
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or signature on informed consent

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
positive seroconversion rate of JE neutralizing antibody following primary vaccination | 28 days after primary vaccination
  to evaluate the positive seroconversion rate of JE neutralizing antibody 28 days after primary vaccination
incidence of solicited adverse reactions (including systemic and local adverse reactions) following primary vaccination | 0-7 days after primary vaccination
  to evaluate incidence of solicited adverse reactions (including systemic and local adverse reactions) within 0-7 days after primary vaccination

SECONDARY OUTCOMES:
GMT of JE neutralizing antibody following primary vaccination | 28 days after primary vaccination
  to evaluate the GMT of JE neutralizing antibody 28 days after primary vaccination
positive seroconversion rate of JE neutralizing antibody following booster vaccination | 28 days after booster vaccination
  to evaluate the positive seroconversion rate of JE neutralizing antibody 28 days after booster vaccination
positive seroconversion rate of JE neutralizing antibody following primary vaccination | 12 months after primary vaccination
  to evaluate the positive seroconversion rate of JE neutralizing antibody 12 months after primary vaccination
incidence of unsolicited adverse reactions (including systemic and local adverse reactions) following primary vaccination | 0-28 days after primary vaccination
  to evaluate incidence of unsolicited adverse reactions (including systemic and local adverse reactions) within 0-28 days after primary vaccination
incidence of adverse event (AE) following booster vaccination | 0-28 days after booster vaccination
  to evaluate incidence of adverse event (AE) within 0-28 days after booster vaccination
incidence of serious adverse event (SAE) during the whole study period | Day 0 of the first dose up to Day 28 of the third dose
  to evaluate incidence of serious adverse event (SAE) during the whole study period
GMT of JE neutralizing antibody following booster vaccination | 28 days after booster vaccination
  to evaluate the GMT and GMI of JE neutralizing antibody 28 days after booster vaccination
GMT of JE neutralizing antibody following primary vaccination | 12 months after primary vaccination
  to evaluate the GMT of JE neutralizing antibody 12 months after primary vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Pizhou Center for Disease Control and Prevention, Xuzhou, Jiangsu, China